CLINICAL TRIAL: NCT01818154
Title: Validation of a New Hand Held Light Emitting Diode (LED) Device for the Determination of Minimal Erythema Dose (MED) for Narrowband Ultraviolet B.
Brief Title: Validation of a New Hand Held Light Emitting Diode Device for the Determination of Minimal Erythema Dose (MED)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study did not start
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Iltefat Hamzavi, Senior Staff Physician, Henry Ford Health System
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 7257
Record Dates: First submitted 2013-03-20; First posted 2013-03-26 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Phototherapy
Keywords: phototherapy; light emitting diode; minimal erythema dose; narrowband UVB

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minimal Erythema Dose LED (Experimental): A 2 x 2 cm section of skin will be exposed to LED light.
  Interventions: Other: LED phototherapy; Other: narrowband UVB phototherapy
- Minimal Erythema Dose narrow band UVB (Placebo Comparator): A 2 x 2 cm section of skin will be exposed to narrow band UVB light.
  Interventions: Other: LED phototherapy; Other: narrowband UVB phototherapy

INTERVENTIONS:
Other: LED phototherapy
Other: narrowband UVB phototherapy

SUMMARY:
The purpose of this study is to validate a new hand held light emitting diode (LED) device for the measurement of minimal erythema dose (MED) for narrow band Ultraviolet B (UVB) radiation by comparing to the traditional approach of measurement of the minimal erythema dose.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years.

Exclusion Criteria:

1. Pregnancy
2. Lactation
3. History of photosensitivity disorder
4. Photosensitizing medications
5. Personal history of melanoma or non-melanoma skin cancer.
6. Skin disease on the back

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Minimal Erythema Dose | 1 day
  The Investigator will look at area irradiated and evaluate for erythema. The lowest dose at which erythema is noted will be recorded as the minimal erythema dose.

CONTACTS AND LOCATIONS:
Overall Officials: Iltefat H Hamzavi, M.D., Principal Investigator — Henry Ford Dermatology
Locations (1):
- Henry Ford Medical Center Department of Dermatology, Detroit, Michigan, United States